CLINICAL TRIAL: NCT01305772
Title: Identification of a Gene Expression Signature Profile for Panitumumab Sensitivity in Untreated Locally Advanced Squamous Cell Cancer of the Head and Neck (SCCHN)
Brief Title: Identification of Gene Expression Signature for Panitumumab Sensitivity in Untreated Locally Advanced SCCHN
Acronym: TOP0901
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated for low accrual.
Sponsor: Neal Ready (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Neal Ready, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00023859; 20080645 (Other: Previous Protocol ID)
Record Dates: First submitted 2011-02-14; First posted 2011-03-01 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: SCCHN; untreated; Stage III or IVa-b (M0)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Panitumumab; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Experimental): Patients who underwent surgery after research PET/CT scans and subsequent radiation therapy with panitumumab administration
  Interventions: Drug: Panitumumab; Procedure: Surgery; Procedure: Radiation Therapy
- Radiation Therapy (Active Comparator): Patients who underwent radiation therapy only, in conjunction with panitumumab therapy.
  Interventions: Drug: Panitumumab; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Panitumumab — Single dose Panitumumab 9mg/kg IV (in the vein) prior to definitive therapy (surgery or radiation therapy). Two additional doses of panitumumab 9mg/kg IV may be given at weeks 1 & 4 of RT alone or weeks 1 & 4 of cisplatin/RT if they tolerated first dose of panitumumab.
  Other Names: Vectibix®; ABX-EGF
Procedure: Surgery — Second biopsy was taken from surgical resection tissue (when possible obtained pre and post panitumumab biopsies from the same site).
  Arms: Surgery
Procedure: Radiation Therapy — Radiation therapy was initiated within 8 weeks after surgery, or as soon as possible.
  Other Names: RT

SUMMARY:
The purpose of this study was to identify which cancer-related genes are turned on or turned off in order to determine how well a patient will respond to the study drug, panitumumab. Panitumumab was added to standard adjuvant or primary radiation therapy. There were subjects that receive surgery followed by therapy and subjects that receive radiation therapy without surgery.

Subjects entering this study had locally advanced disease that can be treated with surgery and/or radiation therapy. Fresh frozen tumor tissue were available for genomics analysis prior to initiating panitumumab therapy. If fresh frozen tissue was not available at time of consent, a biopsy was required to participate in this trial.

DETAILED DESCRIPTION:
The trial was initiated to identify a gene expression signature profile biomarker for panitumumab sensitivity in locally advanced, untreated SCCHN. SCCHN expresses or over expresses EGFR in >90% of tumors. Panitumumab is a fully human IgG2 monoclonal antibody approved for the treatment of epidermal growth factor receptor (EGFR) expressing previously treated metastatic colorectal cancer. It competes with endogenous ligands such as epidermal growth factor and tumor growth factor-α and blocks stimulation of the EGFR. Preclinical experiments have shown that panitumumab has both direct anti-tumor activity and can activate a cellular immune response to SCCHN.This study provides the opportunity to better define the population of patients that would benefit from EGFR inhibition in SCCHN.

Patients received single agent panitumumab in a "window of opportunity" design prior to definitive surgical or radiation therapy. The decision to treat primarily with either surgery or Radiation Therapy (RT) based therapy was based on best medical practice by the treating physician per National Comprehensive Cancer Network (NCCN) guidelines at www.nccn.org.

Response to panitumumab monotherapy before surgery or radiation was evaluated as a continuous variable, and a median split of patients will be used to develop a signature of drug responsiveness. An Affymetrix chip based gene signature model was then developed by analyzing gene expression in panitumumab sensitive versus resistant tumors. Identification of a gene expression profile for tumor sensitivity allowed for prospective trials treating patient populations enriched for likelihood of clinical benefit from panitumumab therapy. It is also possible that a gene signature profile for panitumumab responsiveness identified in SCCHN could be used as a biomarker in other epithelial cancers.

Tumor response as measured by percentage decrease in PET scan standardized uptake value (SUV) level or objective evidence of tumor response (by CT scan or direct measurement) was the basis for examining the activity of panitumumab by means of identifying a gene expression signature that predicted response in this patient population. Therefore, PET scan SUV levels was assessed at baseline prior to any treatment. If a baseline PET/CT was obtained and a lesion identified with SUV level ≥6, an additional pre-treatment research PET/CT was performed after consent (prior to dose #1 panitumumab. A second research PET/CT was also obtained after the first dose of panitumumab as part of this research study. If no baseline PET/CT had been obtained, a research PET was obtained pre-treatment; if SUV level ≥6 an additional research PET was obtained after the first dose of panitumumab.

All subjects underwent imaging, biopsy and a single dose of panitumumab 9mg/kg IV. Two to three weeks after panitumumab, imaging was repeated and a second biopsy was obtained (at surgery for surgery patients) and an optional biopsy for patients receiving RT. Subjects received 2 additional doses of panitumumab during their standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated, suspected or histologically documented locally advanced clinical stage III or IVa-b(M0)SCCHN, no evidence of distant metastases. Prior surgery with diagnosis of SCCHN acceptable
2. Candidate for definitive surgery or radiation based therapy.
3. Fresh frozen tumor tissue must be available for genomic analysis and must pass RNA Quality Control prior to research PET/CT #1 and/or initiating panitumumab
4. Measurable or evaluable disease
5. Eastern Cooperative Oncology Group (ECOG) 0-1
6. ≥18 years of age
7. Adequate organ function

   1. neutrophil count (ANC or AGC) ≥1.5 x 109/L
   2. Platelet count ≥75 x 109/L
   3. Hemoglobin ≥9.0 g/dL
   4. Creatinine ≤1.5x upper limit of normal (ULN)
   5. Hepatic enzymes (AST, ALT)≤2.5x ULN, Total Bilirubin <1.5x ULN
   6. Magnesium ≥ Lower limit of Normal (LLN)
8. Negative serum pregnancy test ≤7 days before starting panitumumab (for women of childbearing potential only)
9. Competent to comprehend, sign, and date a written informed consent form
10. Sexually active males & females of reproductive potential must agree to use adequate method of contraception during treatment & for 6 months after study drug stopped

Exclusion Criteria:

1. History of other malignancy within past 2 years, except:

   1. Malignancy treated with curative intent and with no known active disease
   2. Adequately treated non-melanomatous skin cancer or lentigo maligna with no evidence of disease
   3. Adequately treated cervical carcinoma in situ with no evidence of disease
   4. Prostatic intraepithelial neoplasia with no evidence of prostate cancer
2. Primary tumor of the nasopharynx (nasopharyngeal cancer), sinuses, salivary gland, or skin. (Squamous cell carcinoma arising in/near nasopharynx is eligible)
3. Prior radiotherapy in planned field if it prevents standard radiotherapy dose and field
4. Prior radiation for head & neck cancer
5. Prior anti-EGFR antibody therapy (e.g., cetuximab) or treatment with small molecule EGFR inhibitors (e.g., gefitinib, erlotinib, lapatinib)
6. Prior anti-cancer treatment with: chemotherapy, hormonal therapy, immunotherapy, experimental or approved proteins/antibodies within the past 5 years.
7. Prior systemic chemotherapy for study cancer
8. Investigational agent or therapy ≤30 days before enrollment and/or have not recovered from such side effects
9. Continued chronic use of immunosuppressive agents during the clinical trial period (e.g., methotrexate and cyclosporine), corticosteroids are allowed
10. Clinically significant cardiovascular disease (including myocardial infarction (MI), unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤6 months before enrollment
11. History of interstitial lung disease e.g., pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan. Patients with CT scan findings consistent with lung scarring from chronic obstructive pulmonary disease (COPD) or previous infection are eligible
12. History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results
13. Unwilling or unable to comply with study requirements
14. Pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
15. Known positive test(s) for HIV infection
16. Major surgery within 2 weeks of enrollment. Staging endoscopy with biopsy/tonsillectomy for head & neck cancer, tracheostomy, and/or gastrostomy tube placement eligible one day after procedure. May consent to tissue collection biopsy pre-endoscopy/minor surgery and then begin protocol therapy one day after procedure.
17. Known allergy/hypersensitivity to any component of the study treatment(s)
18. Infection requiring intravenous antibiotics for any uncontrolled infection ≤14 days prior to enrollment
19. Subjects on anticoagulant therapy. Aspirin and other anti-platelet agents will not be defined as anticoagulant therapy for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients had successful genomic screening and RNA extraction/quality control.
Groups:
- Radiation Therapy: Patients who underwent radiation therapy only, in conjunction with panitumumab therapy.
  Radiation Therapy : Radiation therapy was initiated within 8 weeks after surgery, or as soon as possible.
  Panitumumab : Single dose Panitumumab 9mg/kg IV for a total of 3 doses (if tolerated). Dose #1 is to be administered prior to RT for RT arm. Within the surgery arm, second and third doses of panitumumab were administered after surgery during weeks 1 & 4 of RT. Within the RT arm, second and third doses will be administered at weeks 1 & 4 during RT.
- Surgery: Patients who underwent surgery after research PET/CT scans and subsequent radiation therapy with panitumumab administration
  Panitumumab : Single dose Panitumumab 9mg/kg IV for a total of 3 doses (if tolerated). Dose #1 is to be administered prior to RT for RT arm. Within the surgery arm, second and third doses of panitumumab were administered after surgery during weeks 1 & 4 of RT. Within the RT arm, second and third doses will be administered at weeks 1 & 4 during RT.
  Surgery : Second biopsy was taken from surgical resection tissue (when possible obtained pre and post panitumumab biopsies from the same site).
Period: Overall Study
Arm/Group | Radiation Therapy | Surgery
Started | 5 | 1
Genomic Screening + Biopsy #1 | 5 | 1
Research PET/CT #1 | 5 | 1
Panitumumab Dose #1 | 5 | 1
Research PET/CT #2 | 5 | 1
Surgery/Biopsy #2 | 1 (2nd research tissue sample not collected for 4 patients due to safety risk to subject.) | 1
RT + Panitumumab Dose #2 / #3 | 5 (RT and doses #2 and #3 of panitumumab administered to patients regardless of 2nd biopsy status.) | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy | Surgery | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.60 (6.66) | 69 (NA) — Cannot measure uncertainty about one (1) subject. | 65.33 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor (Primary Tumor and Lymph Node) Response and Progression Between Pre- and Post- Panitumumab Therapy
Description: The aim of this outcome measure was to identify a gene expression signature that predicts response to panitumumab in untreated locally advanced squamous cell cancer of the head / neck (SCCHN). Response and progression were evaluated using the largest percentage change among the cases: 1) Pre-panitumumab PET scan activity, and/or; 2) Pre-panitumumab radiologic measurement compared to post-panitumumab measurement and/or; 3) Pre-panitumumab direct measurement of tumor / lymph node compared to post-panitumumab direct measurement of tumor / lymph node. Response and progression were evaluated in this single study using the criteria "changes in only the largest diameter (unidimensional measurement) of the tumor lesions were defined" in the same manner as in RECIST 1.1.
  No results are reported as only 2 of the 6 subjects had fresh tissue collected after the first dose of panitumumab. The study was amended to remove the biopsy procedure due to the potential risk for the participants.
Time Frame: Baseline to 2 years
Population: No results will be reported for the primary outcome measure as only 2 of the 6 subjects had tissue collected after the first dose of panitumumab due to safety risk to the subject.
Groups:
- Overall Study: Patients from both the Surgery and RT arms will be combined in reporting primary and secondary outcome results, as one arm only contains 1 subject. Statistical uncertainty cannot be measured about 1 subject.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

2. Secondary Outcome: Nine (9) Month Progression Free Survival (PFS)
Description: Nine month progression-free survival (PFS) was defined from the time from enrollment to the first date of disease progression or death as a result of any cause. Progression was defined in the same manner as in RECIST 1.1: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5mm (the appearance of one or more new lesions is also considered progression).
  Time was censored at the date of the last follow-up visit for subjects who were still alive and have not progressed. The 9 month PFS rate is a percentage, representing the fraction of treated subjects who, after 9 months, are disease free or alive.
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: percentage of treated patients
Arm/Group | Overall Study
Number analyzed (Participants) | 6
percentage of treated patients | 60 [12.57 to 88.18]

3. Secondary Outcome: Nine (9) Month Overall Survival (OS)
Description: Overall survival (OS) was defined as from the time of enrollment to the date of death resulting from any cause. Time as censored at the date of the last follow-up visit for subjects who were still alive. The 9-month OS rate is a percentage, representing the fraction of treated subjects who, after 9 months, are alive.
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: percentage of treated patients surviving
Arm/Group | Overall Study
Number analyzed (Participants) | 6
percentage of treated patients surviving | 80 [20.38 to 96.92]

ADVERSE EVENTS:
Groups:
- Radiation Therapy: Radiation therapy with panitumumab therapy.
- Surgery: Surgery after research PET/CT scans and subsequent radiation therapy with panitumumab therapy.
Arm/Group | Radiation Therapy | Surgery
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=5) | Surgery (N=1)
Anemia (Blood and lymphatic system disorders) | 4 | 0
Blood and lymphatic system disorders - Other, specify: Granulocytes (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Eye disorders - Other, specify: Eye Itching (Eye disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Esophageal pain (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify: Odonyphagia (Gastrointestinal disorders) | 5 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Chills (General disorders) | 1 | 1
Edema face (General disorders) | 1 | 1
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 1
Fever (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Gum infection (Infections and infestations) | 3 | 0
Infections and infestations - Other, specify: Face (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 3 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 2 | 1
Weight loss (Investigations) | 5 | 1
White blood cell decreased (Investigations) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: Muscle weakness - Area N/A (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: Mood alteration - Type N/A (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify: Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No